CLINICAL TRIAL: NCT02631577
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Atezolizumab in Combination With Obinutuzumab Plus Lenalidomide in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: A Study Evaluating the Safety and Efficacy of Atezolizumab in Combination With Obinutuzumab Plus Lenalidomide in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29562; 2015-002467-42 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — atezolizumab; Lenalidomide; obinutuzumab

ARMS (2):
- Atezolizumab-G-lena 15mg (Experimental): Participants were administered obinutuzumab, Atezolizumab, and 15 mg of Lenalidomide.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ]; Drug: Lenalidomide; Drug: Obinutuzumab
- Atezolizumab-G-lena 20mg (Experimental): Participants were administered obinutuzumab, Atezolizumab, and 20 mg of Lenalidomide.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ]; Drug: Lenalidomide; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A) [TECENTRIQ] — Atezolizumab will be administered at a flat dose of 840 mg on Days 1 and 15 of Cycles 2 to 6, given in 28-day cycles as induction treatment and 840 mg on Days 1 and 2 of each month, given as maintenance treatment.
Drug: Lenalidomide — Lenalidomide will be administered orally once daily on Days 1 to 21 of Cycles 1 to 6 (28-day cycles) during induction treatment and on Days 1 to 21 of each month during maintenance treatment. Lenalidomide will be administered at a dose of 15 or 20 mg (dose may be de-escalated to 10 mg) during induction treatment and at 10 mg during maintenance treatment. During the expansion phase, lenalidomide will be administered at the RP2D during induction treatment and at 10 mg during maintenance treatment.
Drug: Obinutuzumab — Obinutuzumab will be administered by intravenous infusion at an absolute (flat) dose of 1000 mg on Days 1, 8, and 15 of the first cycle and on Day 1 of each subsequent cycle during induction treatment, and on Day 1 of every other month (i.e., every 2 months) during maintenance treatment.

SUMMARY:
This study will evaluate the safety, efficacy, pharmacokinetics and immunogenicity of induction treatment consisting of atezolizumab in combination with obinutuzumab plus lenalidomide in patients with relapsed or refractory follicular lymphoma (FL), followed by maintenance treatment with atezolizumab plus obinutzumab plus lenalidomide in patients who achieve a complete response (CR), a partial response (PR), or stable disease at end of induction.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Relapsed or refractory FL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody and for which no other more appropriate treatment option exists as determined by the investigator
* Histologically documented CD20-positive lymphoma as determined by the local laboratory
* Fluorodeoxyglucose-avid lymphoma (i.e., PET-positive lymphoma)
* At least one bi-dimensionally measurable lesion (>1.5 cm in its largest dimension by CT scan or magnetic resonance imaging [MRI])
* Availability of a representative tumor specimen and the corresponding pathology report for retrospective central confirmation of the diagnosis of FL
* Agreement to comply with all local requirements of the lenalidomide risk minimization plan
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period (including periods of treatment interruption), and for at least 18 months after the last dose of study treatment
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm for at least 3 months after the last dose of study treatment

Exclusion Criteria:

* Grade 3b follicular lymphoma
* History of transformation of indolent disease to diffuse large B-cell lymphoma (DLBCL)
* Known CD20-negative status at relapse or progression
* Central nervous system lymphoma or leptomeningeal infiltration
* Prior allogeneic stem-cell transplantation (SCT)
* Completion of autologous SCT within 100 days prior to Day (D) 1 of Cycle (C) 1
* Prior standard or investigational anti-cancer therapy as specified in protocol
* History of resistance to lenalidomide or response duration of <1 year
* Treatment with systemic immunosuppressive medications
* History of solid organ transplantation
* Clinically significant toxicity from prior therapy that has not resolved to Grade <=2 (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE], v4.0) prior to Day 1 of Cycle 1
* History of erythema multiforme, Grade >= 3 rash, or blistering following prior treatment with immunomodulatory derivatives such as thalidomide and lenalidomide
* Active bacterial, viral, fungal, or other infection
* Positive for hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody at screening
* Known history of HIV positive status
* History of progressive multifocal leukoencephalopathy
* History of autoimmune disease
* Contraindication to treatment for TE prophylaxis
* Grade <= 2 neuropathy
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of any significant, uncontrolled concomitant disease
* Inadequate hematologic function (unless due to underlying lymphoma)
* Abnormal laboratory values (unless due to underlying lymphoma)
* Pregnant or lactating or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University Miami, Miami, Florida
  - Norton Medical Plaza II, Louisville, Kentucky
  - Memorial Sloan-Kettering Cancer Center; Hematology/Oncology, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
- France (11):
  - Chu Toulouse, Bron
  - Hopital Henri Mondor; 51 Av Mal Lattre De Tassigny, Créteil
  - Hopital du Bocage, Dijon
  - Centre Jean Bernard, Le Mans
  - Centre Hospitalier Le Mans, Le Mans
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - CHU Montpellier - Saint ELOI, Montpellier
  - CHU - Hôtel Dieu hematolgie clinique, Nantes
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - Centre Henri Becquerel, Rouen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in France (9) and USA (5).
Pre-assignment Details: All participants received daily low-dose aspirin (81-100 mg) during lenalidomide treatment and until 28 days after the last dose of lenalidomide. Participants who are unable to tolerate aspirin, who have a history of thromboembolism (TE), and who are at high risk of TE, received warfarin or low-molecular-weight heparin (LMWH).
Period: Overall Study
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Started | 4 | 34
Completed | 3 | 24
Not Completed | 1 | 10
Not completed — Death | 1 | 7
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg | Total
Number analyzed (Participants) | 4 | 34 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (9.1) | 60.4 (9.7) | 60.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 18 | 19
  Male | 3 | 16 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 13 | 16
  Not Stated | 0 | 12 | 12
  Unknown | 0 | 9 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Unknown | 0 | 20 | 20
  White | 4 | 14 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) at End of Induction (EOI), as Determined by the Independent Review Committee (IRC) Using Modified Lugano 2014 Criteria
Description: Complete response (CR) was evaluated through use of PET-CT scans, using the Modified Lugano 2014 criteria. Response was determined by the IRC.
Time Frame: 6 months (up to clinical cut-off date (CCOD) of 23 October 2018)
Population: As no DLTs were observed, the dose of 20 mg lenalidomide was confirmed as the recommended Phase II dose (RP2D) for lenalidomide. Only participants who received lenalidomide induction at the 20 mg RP2D were included in the Efficacy Evaluable population, hence participants in the Atezo-G-L 15 mg arm were not included in the efficacy analysis.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage of Participants |  | 71.9 [56.06 to 84.47]

2. Secondary Outcome: Percentage of Participants Achieving CR at EOI, as Determined by the Investigator Using Modified Lugano 2014 Criteria
Description: CR was evaluated through use of PET-CT scans, using the Modified Lugano 2014 criteria. Response was determined by the Investigator.
Time Frame: 6 months (up to CCOD of 23 October 2018)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage of Participants |  | 75 [59.39 to 86.91]

3. Secondary Outcome: Percentage of Participants Achieving CR at EOI, as Determined by the IRC and Investigator Using Lugano 2014 Criteria
Description: CR was evaluated through use of CT scans, using the Lugano 2014 criteria. Response was determined by the IRC and by the Investigator.
Time Frame: 6 months (up to CCOD of 23 October 2018)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage of Participants
  Determined by the IRC with CT or MRI |  | 31.3 [18.04 to 47.21]
  Determined by Investigator with CT or MRI |  | 50 [34.41 to 65.59]

4. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI as Determined by the IRC and Investigator on the Basis of PET-CT Scans
Description: Objective response was evaluated through use of PET-CT scans, using the Lugano 2014 or modified Lugano 2014 criteria. Response was determined by the IRC and by the Investigator.
Time Frame: 6 months (up to CCOD of 23 October 2018)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage of Participants
  Determined by IRC, based on Lugano 2014 - PET |  | 81.3 [66.31 to 91.50]
  Determined by Inv., based on Lugano 2014 - PET |  | 84.4 [69.92 to 93.63]
  Determined by IRC, Modified Lugano 2014 - PET-CT |  | 78.1 [62.81 to 89.26]
  Determined by Inv, Modified Lugano 2014 - PET-CT |  | 84.4 [69.92 to 93.63]

5. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI as Determined by the IRC and Investigator on the Basis of CT Scans Alone
Description: Objective response was evaluated through use of CT scans alone, using the Lugano 2014. Response was determined by the IRC and by the Investigator.
Time Frame: 6 months (up to CCOD of 23 October 2018)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage of Participants
  Determined by IRC, based on Lugano 2014 - CT |  | 81.3 [66.31 to 91.50]
  Determined by Inv., based on Lugano 2014 - CT |  | 87.5 [73.64 to 95.62]

6. Secondary Outcome: Percentage of Participants With Best Response (CR or PR) During the Study as Determined by the Investigator on the Basis of CT Scans Alone
Description: Best Response was evaluated through use of CT scans alone, using the Lugano 2014. Response was determined by the Investigator.
Time Frame: 30 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 0 | 32
Percentage
  Best Response (CR,PR) |  | 87.5 [73.64 to 95.62]
  CR |  | 68.8 [52.79 to 81.96]
  PR |  | 18.8 [8.50 to 33.69]

7. Secondary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
Participants
  Adverse Events | 4 | 34
  Serious Adverse Events | 2 | 16

8. Secondary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) During Cycle 2 of Study Treatment
Description: Does limiting toxicity (DLT) is defined as any one of the following events occurring during Cycle 2 of treatment and assessed by the investigator as related to study treatment: - Adverse event of any grade that leads to a delay of more than 14 days at the start of the next treatment cycle; - Hematologic adverse events (neutropenia, thrombocytopenia); - Non-hematologic adverse event, except IRRs, diarrhea, nausea or vomiting
Time Frame: Day 1 - Day 28 of second cycle
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
Number of Participants | 0 | 0

9. Secondary Outcome: Serum Concentration of Obinutuzumab (mcg/mL)
Description: The following abbreviations apply in the table: Ind C = Induction Cycle; D = Day; Maint M = Maintenance Month; TRTC = Study Drug Completion or Early Discontinuation; PK FU = Pharmacokinetics and Immunogenicity Follow-up; YR = Year
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
mcg/mL
  Ind C1 D1 - Predose: number analyzed (Participants) | 0 | 2
  Ind C1 D1 - Predose |  | 0.634 (0.857)
  Ind C1 D1 - 30 min. Postdose: number analyzed (Participants) | 4 | 30
  Ind C1 D1 - 30 min. Postdose | 364 (45.9) | 375 (163)
  Ind C2 D1 - Predose: number analyzed (Participants) | 4 | 32
  Ind C2 D1 - Predose | 288 (84.2) | 392 (164)
  Ind C2 D1 - 30 min. Postdose: number analyzed (Participants) | 4 | 31
  Ind C2 D1 - 30 min. Postdose | 606 (62.4) | 753 (225)
  Ind C4 D1 - Predose: number analyzed (Participants) | 3 | 25
  Ind C4 D1 - Predose | 175 (38.5) | 301 (150)
  Ind C4 D1 - 30 min. Postdose: number analyzed (Participants) | 3 | 23
  Ind C4 D1 - 30 min. Postdose | 509 (47.0) | 657 (198)
  Ind C6 D1 - Predose: number analyzed (Participants) | 3 | 20
  Ind C6 D1 - Predose | 230 (12.3) | 272 (106)
  Ind C6 D1 - 30 min. Postdose: number analyzed (Participants) | 3 | 20
  Ind C6 D1 - 30 min. Postdose | 503 (25.5) | 652 (177)
  Maint M1 - Predose: number analyzed (Participants) | 3 | 20
  Maint M1 - Predose | 114 (16.7) | 201 (104)
  Maint M7 - Predose: number analyzed (Participants) | 2 | 17
  Maint M7 - Predose | 66.1 (20.4) | 112 (52.1)
  Maint M13 - Predose: number analyzed (Participants) | 1 | 18
  Maint M13 - Predose | 77.9 (NA) — The standard deviation couldn't be calculated from one participant. | 104 (62.9)
  Maint M19 - Predose: number analyzed (Participants) | 2 | 12
  Maint M19 - Predose | 94.0 (24.0) | 111 (49.8)
  TRTC: number analyzed (Participants) | 0 | 12
  TRTC |  | 148 (103)
  OD120FU: number analyzed (Participants) | 1 | 10
  OD120FU | 23.3 (NA) — The standard deviation couldn't be calculated from one participant. | 46.2 (38.6)
  O1YFU: number analyzed (Participants) | 2 | 4
  O1YFU | 46.9 (66.2) | 57.9 (115)

10. Secondary Outcome: Serum Concentration of Atezolizumab (mcg/mL)
Description: as for outcome 9
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
micrograms per milliliter (mcg/mL)
  Ind C2 D1 - Predose: number analyzed (Participants) | 0 | 1
  Ind C2 D1 - Predose |  | 0.184 (NA) — The standard deviation couldn't be calculated from one participant.
  Ind C2 D1 - 30 min. Postdose: number analyzed (Participants) | 4 | 32
  Ind C2 D1 - 30 min. Postdose | 345 (195) | 279 (123)
  Ind C2 D15 - Predose: number analyzed (Participants) | 3 | 32
  Ind C2 D15 - Predose | 73.8 (6.47) | 90.0 (33.8)
  Ind C4 D1 - Predose: number analyzed (Participants) | 2 | 29
  Ind C4 D1 - Predose | 128 (33.9) | 226 (93.9)
  Ind C4 D1 - 30 min. Postdose: number analyzed (Participants) | 2 | 27
  Ind C4 D1 - 30 min. Postdose | 340 (38.2) | 477 (126)
  Ind C6 D1 - Predose: number analyzed (Participants) | 3 | 28
  Ind C6 D1 - Predose | 194 (40.6) | 279 (117)
  Maint M1 - Predose: number analyzed (Participants) | 3 | 27
  Maint M1 - Predose | 79.0 (67.6) | 172 (76.5)
  Maint M1 - Day 2, 30 min. Postdose: number analyzed (Participants) | 3 | 23
  Maint M1 - Day 2, 30 min. Postdose | 653 (106) | 666 (185)
  Maint M4 - Predose: number analyzed (Participants) | 3 | 25
  Maint M4 - Predose | 174 (32.9) | 292 (97.1)
  Maint M7 - Predose: number analyzed (Participants) | 2 | 20
  Maint M7 - Predose | 209 (12.7) | 322 (109)
  Maint M13 - Predose: number analyzed (Participants) | 1 | 19
  Maint M13 - Predose | 203 (NA) — The standard deviation couldn't be calculated from one participant. | 309 (140)
  Maint M19 - Predose: number analyzed (Participants) | 1 | 11
  Maint M19 - Predose | 351 (NA) — The standard deviation couldn't be calculated from one participant. | 327 (140)
  TRTC: number analyzed (Participants) | 0 | 13
  TRTC |  | 116 (81.9)
  PK FU 120D: number analyzed (Participants) | 1 | 11
  PK FU 120D | 46.0 (NA) — The standard deviation couldn't be calculated from one participant. | 38.4 (24.6)
  PK FU 1YR: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Serum Concentration of Lenalidomide (ng/mL)
Description: The following abbreviations apply in the table: Ind C = Induction Cycle; D = Day; HR = Hour
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
nanograms/milliliter (ng/mL)
  Ind C1 D1 - Predose: number analyzed (Participants) | 0 | 0
  Ind C1 D15 - Predose: number analyzed (Participants) | 4 | 17
  Ind C1 D15 - Predose | 12.6 (14.3) | 13.0 (11.4)
  Ind C1 D15 - 2.0 hr. Postdose: number analyzed (Participants) | 4 | 18
  Ind C1 D15 - 2.0 hr. Postdose | 254 (115) | 294 (114)
  Ind C2 D15 - Predose: number analyzed (Participants) | 3 | 21
  Ind C2 D15 - Predose | 3.57 (3.25) | 15.0 (13.0)
  Ind C2 D15 - 30 min. Postdose: number analyzed (Participants) | 3 | 19
  Ind C2 D15 - 30 min. Postdose | 241 (116) | 293 (233)
  Ind C2 D15 -1.0 hr. Postdose: number analyzed (Participants) | 3 | 20
  Ind C2 D15 -1.0 hr. Postdose | 224 (43.1) | 354 (120)
  Ind C2 D15 - 2.0 hr. Postdose: number analyzed (Participants) | 3 | 19
  Ind C2 D15 - 2.0 hr. Postdose | 146 (41.9) | 262 (82.1)
  Ind C2 D15 - 4.0 hr. Postdose: number analyzed (Participants) | 3 | 20
  Ind C2 D15 - 4.0 hr. Postdose | 95.8 (18.3) | 150 (47.1)
  Ind C2 D15 - 8.0 hr. Postdose: number analyzed (Participants) | 3 | 20
  Ind C2 D15 - 8.0 hr. Postdose | 45.9 (23.9) | 68.4 (33.6)
  Ind C6 D15 - Predose: number analyzed (Participants) | 3 | 12
  Ind C6 D15 - Predose | 5.72 (3.73) | 9.17 (6.87)
  Ind C6 D15 - 2.0 hr. Postdose: number analyzed (Participants) | 3 | 12
  Ind C6 D15 - 2.0 hr. Postdose | 200 (57.5) | 214 (77.6)

12. Secondary Outcome: Number of Participants Positive for Human Anti-human Antibodies (HAHA) to Obinutuzumab
Description: The following abbreviations apply in the table: Ind C = Induction Cycle; D = Day; Maint M = Maintenance Month; TRTC = Study Drug Completion or Early Discontinuation; PK FU = Pharmacokinetics and Immunogenicity Follow-up; YR = Year. All baseline and post-baseline samples from participants were negative for HAHAs to obinutuzumab and the results are shown below.
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
Participants
  Baseline - Negative | 4 | 34
  Ind C6 D1 - Negative: number analyzed (Participants) | 3 | 27
  Ind C6 D1 - Negative | 3 | 27
  Study drug completion or early discontinuation - Negative: number analyzed (Participants) | 0 | 15
  Study drug completion or early discontinuation - Negative | 0 | 15
  OB, PK, IMMUNO FU 120D - Negative: number analyzed (Participants) | 1 | 11
  OB, PK, IMMUNO FU 120D - Negative | 1 | 11
  OB, PK, IMMUNO FU 1YR - Negative: number analyzed (Participants) | 2 | 4
  OB, PK, IMMUNO FU 1YR - Negative | 2 | 4

13. Secondary Outcome: Number of Participants Positive for Anti-therapeutic Antibodies (ATAs) to Atezolizumab
Description: The following abbreviations apply in the table: Ind C = Induction Cycle; D = Day; Maint M = Maintenance Month; TRTC = Study Drug Completion or Early Discontinuation; PK FU = Pharmacokinetics and Immunogenicity Follow-up; YR = Year. All baseline and post-baseline samples were negative for ATAs to atezolizumab and the results are shown below.
Time Frame: Baseline up to approximately 59 months
Population: The Safety Evaluable Population included participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
Number analyzed (Participants) | 4 | 34
Participants
  Ind C2 D1 - Negative: number analyzed (Participants) | 4 | 31
  Ind C2 D1 - Negative | 4 | 31
  Ind C2 D15 - Negative: number analyzed (Participants) | 2 | 32
  Ind C2 D15 - Negative | 2 | 32
  Ind C4 D1 - Negative: number analyzed (Participants) | 3 | 29
  Ind C4 D1 - Negative | 3 | 29
  Ind C6 D1 - Negative: number analyzed (Participants) | 3 | 28
  Ind C6 D1 - Negative | 3 | 28
  Maint M1 - Negative: number analyzed (Participants) | 3 | 27
  Maint M1 - Negative | 3 | 27
  Maint M4 - Negative: number analyzed (Participants) | 3 | 25
  Maint M4 - Negative | 3 | 25
  Maint M7 - Negative: number analyzed (Participants) | 2 | 21
  Maint M7 - Negative | 2 | 21
  Maint M13 - Negative: number analyzed (Participants) | 1 | 20
  Maint M13 - Negative | 1 | 20
  Maint M19 - Negative: number analyzed (Participants) | 2 | 12
  Maint M19 - Negative | 2 | 12
  Study drug completion or early discontinuation - Negative: number analyzed (Participants) | 2 | 15
  Study drug completion or early discontinuation - Negative | 2 | 15
  ATEZO, PK, IMMUNO FU 120D - Negative: number analyzed (Participants) | 1 | 11
  ATEZO, PK, IMMUNO FU 120D - Negative | 1 | 11
  ATEZO, PK, IMMUNO FU 1YR - Negative: number analyzed (Participants) | 2 | 3
  ATEZO, PK, IMMUNO FU 1YR - Negative | 2 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 59 months
Description: The safety population included all participants who received at least one treatment with study medication. The adverse event severity grading scale for the NCI CTCAE v4.0 was used.
Arm/Group | Atezolizumab-G-lena 15mg | Atezolizumab-G-lena 20mg
All-Cause Mortality (participants affected / at risk) | 1/4 | 7/34
Serious Adverse Events (participants affected / at risk) | 2/4 | 16/34
Other Adverse Events (participants affected / at risk) | 4/4 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab-G-lena 15mg (N=4) | Atezolizumab-G-lena 20mg (N=34)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0)
ADMINISTRATION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ATYPICAL FIBROXANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SARCOMATOID CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab-G-lena 15mg (N=4) | Atezolizumab-G-lena 20mg (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (4) | 14 (43)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 9 (14)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (2)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 7 (9)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 6 (6)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 8 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (3) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 3 (5) | 12 (13)
DIARRHOEA (Gastrointestinal disorders) | 3 (9) | 19 (42)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 3 (6)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 4 (7)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (8) | 3 (4)
ASTHENIA (General disorders) | 0 (0) | 14 (20)
AXILLARY PAIN (General disorders) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 8 (10)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (2) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 5 (8)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 3 (3) | 5 (6)
XEROSIS (General disorders) | 0 (0) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 0 (0) | 3 (4)
BRONCHIOLITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 10 (13)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 2 (2)
FUNGAL SKIN INFECTION (Infections and infestations) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 6 (10)
PHARYNGITIS (Infections and infestations) | 0 (0) | 3 (3)
RHINITIS (Infections and infestations) | 0 (0) | 9 (12)
SINUSITIS (Infections and infestations) | 4 (5) | 7 (13)
TINEA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 5 (8)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (4)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (2) | 11 (12)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 2 (2)
AMYLASE INCREASED (Investigations) | 1 (2) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2)
LIPASE INCREASED (Investigations) | 1 (2) | 4 (6)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (10)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (15)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (4)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 2 (3)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 4 (4)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 2 (2) | 2 (2)
INSOMNIA (Psychiatric disorders) | 1 (1) | 4 (5)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 12 (14)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 2 (2)
DRY EYE (Eye disorders) | 0 (0) | 2 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 4 (6)
MALAISE (General disorders) | 0 (0) | 2 (2)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 2 (2)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 2 (2)
CYSTITIS (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 5 (5)
DYSURIA (Renal and urinary disorders) | 0 (0) | 3 (3)
HOT FLUSH (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment for this study was stopped early as the Sponsor chose not to claim superiority over existing therapies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02631577/Prot_SAP_001.pdf